CLINICAL TRIAL: NCT07357493
Title: The CARBO Study (metaCARpal Bone Osteosynthesis)
Brief Title: metaCARpal Bone Osteosynthesis Trail
Acronym: CARBO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University (Other); Umeå University (Other); University of Oslo (Other); Tampere University (Other); Københavns Universitet (Other); Göteborg University (Other); Linkoeping University (Other Government); Region Stockholm (Other Government); Östersund Hospital (Unknown)
Responsible Party: Principal Investigator, Cecilia Mellstrand Navarro, MD PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-04413-01; FoUI-1022484 (Other Grant/Funding Number: ALF Region Stockholm)
Record Dates: First submitted 2025-12-15; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Metacarpal Shaft Fractures
Keywords: Non-operative; operative; metacarpal; shaft; displaced; mobilization
MeSH Terms: interventions — Early Ambulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-operative with early mobilization (Experimental): Participants randomized to the nonoperative group will receive immediate unrestricted mobilization, with optional buddy taping or removable splinting for comfort. Closed reduction will not be attempted. Rehabilitation protocol with early mobilization will be standardized across study centers with printed standardized information to patients and rehabilitation staff.
  Interventions: Procedure: Non-operative treatment with early mobilization
- Operative (Active Comparator): Participants randomized to the operative group will undergo open reduction and internal fixation (ORIF) of the MSF. Peri-operative antibiotic prophylaxis will be administered according to local guidelines. The surgical approach and fixation method (e.g. compression screws and/or plate, not K-wires) will be at the discretion of the treating surgeon, following standard surgical principles. Postoperative immobilisation will adhere to surgeons' preference but not exceed two weeks fixation.
  Interventions: Procedure: Operative treatment

INTERVENTIONS:
Procedure: Non-operative treatment with early mobilization — Participants randomized to the nonoperative group will receive immediate unrestricted mobilization, with optional buddy taping or removable splinting for comfort. Closed reduction will not be attempted. Rehabilitation protocol with early mobilization will be standardized across study centers with printed standardized information to patients and rehabilitation staff.
  Arms: Non-operative with early mobilization
Procedure: Operative treatment — Participants randomized to the operative group will undergo open reduction and internal fixation (ORIF) of the MSF. Peri-operative antibiotic prophylaxis will be administered according to local guidelines. The surgical approach and fixation method (e.g. compression screws and/or plate, not K-wires) will be at the discretion of the treating surgeon, following standard surgical principles. Postoperative immobilisation will adhere to surgeons' preference but not exceed two weeks fixation.
  Arms: Operative

SUMMARY:
Background Metacarpal shaft fractures account for 30-50% of hand fractures (Karl et al., 2015; Kollitz et al., 2014; van Onselen et al., 2003), with diaphyseal spiral and oblique fractures of the second to fifth ray posing unique challenges due to the risks of shortening and rotational deformities. Current standard care of displaced fractures involves operative fixation.

However, retrospective studies have indicated that nonoperative treatment, involving early mobilization or buddy taping, can achieve outcomes comparable to operative treatment (Daher et al., 2023). There is only one published, with a small sample size, randomized controlled trial (RCT) investigating this issue (Peyronson et al., 2023). This highlights the need for a robust multicenter RCT to address these gaps in evidence.

Aim The aim of this study is to compare the one-year outcomes of non-operative treatment involving immediate unrestricted mobilization versus operative treatment of displaced oblique or spiral diaphyseal metacarpal fractures in adults.

Materials and Methods This is a multicenter, pragmatic, prospective, noninferiority RCT involving 552 adult patients with displaced oblique and/or spiral diaphyseal metacarpal fractures of the second to fifth ray. Participants will be randomized 1:1 to receive either nonoperative treatment with unrestricted mobilization and rehabilitation) or operative treatment (with screw or plate fixation) followed by rehabilitation.

The primary outcome is grip-strength in the injured hand presented in kilograms at one year.

Secondary outcomes include questionnaires, complications, range of motion, patient reported outcome measures, health related quality of life, patient satisfaction, and radiographic healing.

A power calculation proposes a study size of 552 participants to detect a noninferiority margin of 10% in grip strength.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Single, displaced spiral or oblique diaphyseal fracture of the second to fifth metacarpals with definition of diaphysis as described by AO 2018 (AO/OTA as 77.2-5.2A) (Meinberg et al., 2018).
* Fracture line length at least twice the diameter of the bone at the level of the fracture (figure 1).
* Fractures with at least 2 mm of radiological displacement and/or malrotation of injured finger compared to uninjured side regardless of fracture displacement.
* Injury within 10 days prior to inclusion.
* Normal bilateral hand function prior to injury.

Exclusion Criteria:

* Presence of contaminated wounds with need for surgical debridement.
* Generalized degenerative joint condition.
* Prior injury to the hand with remaining disability.
* Dementia or other severe cognitive dysfunction.
* Language barrier impeding understanding of study purpose or questionnaires.
* Substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2030-03-15 (Estimated); Study Completion 2031-03-15 (Estimated)

PRIMARY OUTCOMES:
Grip strength | From enrollment to the end of follow-up at 12 months
  The primary outcome is grip-strength measured in the injured hand using a JAMAR dynamometer at 12 months and presented in kilograms. Measurement method will follow the technical description presented in the HAKIR manual (HAKIR, 2023).

SECONDARY OUTCOMES:
Complications | From enrollment to the end of follow-up at 12 months
  infection, malunion, nerve injury, reoperation
Pain in injured hand NRS | From enrollment to the end of follow-up at 12 months
  NRS (Numerical Rating Scale) at rest and when it is at its worst
Rotational deformity | 12 months
  0 - no deformity, 1 - minimal deformity, 2 - clearly visible deformity but acceptable functional limitation, 3 - great deformity and functional limitation
PROM - patient rated outcome measure | 6, 12 weeks, 12 months
  Quick-DASH-9 score (Gabel et al., 2009)
Range of motion | 6, 12 weeks, 12 months
  total active motion and extension lag
Pinch grip strength | 12 weeks, 12 months
Radiographic shortening | 12 months
  according to Sletten (Sletten et al., 2013)
Radiographic healing | 12 weeks, 12 months
  defined as bridging callus formation over the fracture line on a plain x-ray anterio-posterior and/or lateral projection. (Hayes et al., 2023)
Sick leave duration | 12 months
  in days
Patient satisfaction | From enrollment to the end of follow-up at 12 months
  Patient Acceptable Symptom State, PASS (Daryoush et al., 2025)
Quality of life measured by PROM | From enrollment to the end of follow-up at 12 months
  EQ-5D EuroQol Group, 1990; Taft et al., 2004)
Quality of life measured by SF-12 | From enrollment to the end of follow-up at 12 months
  SF-12 (EuroQol Group, 1990; Taft et al., 2004)

IPD SHARING:
Plan to Share IPD: No
Data on group level will be made available upon reasonable request.